CLINICAL TRIAL: NCT03604198
Title: An Open-Label Extension Study of the Safety of Relacorilant (CORT125134) in the Treatment of the Signs and Symptoms of Endogenous Cushing Syndrome
Brief Title: Extension Study to Evaluate the Safety of Long-Term Use of Relacorilant in Patients With Cushing Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-452
Record Dates: First submitted 2018-05-01; First posted 2018-07-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cushing Syndrome
Keywords: Cushing Syndrome; Cushing Disease; Cushing; Hypercortisolemia; Cushingoid; Type 2 Diabetes; Impaired Glucose Intolerance; Hypertension; Adrenal Corticotrophic Hormone (ACTH); Adrenocortical Carcinoma; Primary Pigmented Nodular Adrenal Disease (PPNAD); Moon Facies; Dorsocervical Fat Pad; Adrenal Adenoma; Adrenal Carcinoma; Adrenal Autonomy; Cortisol
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; ACTH Syndrome, Ectopic; Diabetes Mellitus, Type 2; Hypertension; Adrenocortical Carcinoma; Adrenal Cortex Neoplasms | interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- relacorilant (CORT125134) (Experimental)
  Interventions: Drug: relacorilant

INTERVENTIONS:
Drug: relacorilant — CORT125134 is supplied as capsules for oral dosing.
  Other Names: CORT125134

SUMMARY:
This is an open-label extension study to evaluate the long-term safety of relacorilant in patients with endogenous Cushing syndrome who successfully completed participation in a Corcept-sponsored study of relacorilant and may benefit from continuing treatment.

DETAILED DESCRIPTION:
This study is designed to allow continued therapy with relacorilant, a potent, selective glucocorticoid receptor (GR) antagonist in patients who have successfully completed participation of a Corcept-sponsored study of relacorilant (referred to as the "parent" study). Patients may qualify to enter this extension study if they complete their last treatment visit in their parent study and in the Investigator's opinion will benefit from continued treatment.

Once-daily dosing with relacorilant may continue for patients who receive clinical benefits (as judged by the Investigator) until relacorilant is commercially or otherwise available or the study is stopped by the Sponsor. A patient's dose may be maintained, reduced, or increased based on individual response and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Major Inclusion Criteria:

  * Have completed a Corcept-sponsored study of relacorilant in endogenous Cushing syndrome with at least 80% compliance with the dosing schedule.
  * According to the Investigator's opinion will benefit from continuing treatment with relacorilant

Exclusion Criteria:

* Major Exclusion Criteria:

  * Premature discontinuation from a relacorilant parent study.
  * Has uncontrolled, clinically significant hypothyroidism or hyperthyroidism
  * Has poorly controlled hypertension
  * Has Stage ≥ 4 renal failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of relacorilant | 36 months
  Number of participants with treatment-emergent adverse events (TEAEs)as assessed by CTCAE v4.0

OTHER OUTCOMES:
Long-term benefit of relacorilant | 36 months
  Changes from Baseline as measured by glycated hemoglobin(HbA1c) and insulin resistance in patients with diabetes mellitus (DM) or glucose intolerance at Baseline in the parent study
Long-term benefit of relacorilant | 36 months
  Changes from Baseline as measured by systolic and diastolic blood pressure (BP) by ambulatory BP measurements (ABPM) in patients with uncontrolled hypertension (HTN) at Baseline in the parent study and in patients with controlled HTN taking at least one anti-HTN medication.
Long-term benefit of relacorilant | 36 months
  Changes from Baseline in weight as measured by Kg
Long-term benefit of relacorilant | 36 months
  Changes from Baseline in waist circumference measured in cm
Long-term benefit of relacorilant | 36 months
  Changes from Baselinein quality-of-life based on Cushing quality of life questionnaire 0 (worst) to 100 (best)
Long-term benefit of relacorilant | 36 months
  Changes from Baseline in hypthalamic-pituitary-adrenal (HPA) axis markers (Plasma ACTH and Fasting Cortisol) and Sex steroid hormone (testosterone and estradiol)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ru, MD, PhD, Study Director — Corcept Therapeutics
Locations (48):
- United States (25):
  - Site 49, Phoenix, Arizona
  - Site 35, Stanford, California
  - Site 39, Torrance, California
  - Site 50, Miami, Florida
  - Site 10, Atlanta, Georgia
  - Site 9, Chicago, Illinois
  - Site 1, Indianapolis, Indiana
  - Site 5, Metairie, Louisiana
  - Site 27, Baltimore, Maryland
  - Site 13, Fall River, Massachusetts
  - Site 8, Ann Arbor, Michigan
  - Site 36, Rochester, Minnesota
  - Site 34, Jackson, Mississippi
  - Site 3, St Louis, Missouri
  - Site 55, Reno, Nevada
  - Site 6, Albany, New York
  - Site 24, New York, New York
  - Site 4, Wilmington, North Carolina
  - Site 43, Cleveland, Ohio
  - Site 2, Pittsburgh, Pennsylvania
  - Site 46, Pittsburgh, Pennsylvania
  - Site 11, Dallas, Texas
  - Site 7, El Paso, Texas
  - Site 32, Fort Worth, Texas
  - Site 12, Houston, Texas
- Site 14, Vienna, Austria
- Site 51, Nova Scotia, Canada
- Germany (2):
  - Site 16, Munich
  - Site 42, Würzburg
- Israel (2):
  - Site 20, Ramat Gan
  - Site 29, Tel Aviv
- Italy (6):
  - Site 40, Ancona
  - Site 44, Messina
  - Site 25, Milan
  - Site 21, Napoli
  - Site 48, Padua
  - Site 52, Torino
- Site 33, Rotterdam, Netherlands
- Poland (2):
  - Site 47, Krakow
  - Site 45, Lublin
- Romania (3):
  - Site 37, Bucharest
  - Site 31, Bucharest
  - Site 28, Bucharest
- Spain (5):
  - Site 53, Alicante
  - Site 18, Girona
  - Site 17, Madrid
  - Site 38, Málaga
  - Site 19, Seville

IPD SHARING:
Plan to Share IPD: No